CLINICAL TRIAL: NCT03900195
Title: The Effectiveness of Bottle-PEP in Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 09.2019.052
Record Dates: First submitted 2019-01-20; First posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bottle PEP (Experimental): Bottle PEP is a positive expiratory system that is applied via a tube of more than 5 mm of thickness and a bottle filled with water about 10 cms.
  Interventions: Other: BottlePEP
- Control (No Intervention): No interventions will be applied.

INTERVENTIONS:
Other: BottlePEP — Positive expiratory device with a bottle
  Arms: Bottle PEP

SUMMARY:
The effectiveness of Bottle PEP in patients with Chronic Obstructive Pulmonary Disease

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with COPD
* Stable Disease

Exclusion Criteria:

* Neuromuscular disease
* Recent pneumothorax
* Major surgery in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-01-21 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Forced expiratory volume in the first minute | 6 months after intervention
  Pulmonary function tests that are done with a spirometry to measure forced expiratory volume

SECONDARY OUTCOMES:
6 minute walking test | 6 months after intervention
  6 minute walking test is a field test that measures the distance a patient walks during a 6 minute period.
St. George's Quality of Life Score | 6 months after intervention
  Scores are calculated for three domains:
  Symptoms, Activity and Impacts (Psycho-social) as well as a total score.
  Psychometric testing has demonstrated its repeatability, reliability and validity. Sensitivity has been demonstrated in clinical trials.
  A minimum change in score of 4 units was established as clinically relevant after patient and clinician testing. This score has been used in a range of disease groups including asthma, chronic obstructive pulmonary disease and bronchiectasis, and in a range of settings such as randomised controlled therapy trials and population surveys.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Medicine Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No